CLINICAL TRIAL: NCT02662595
Title: Mimi - mHealth to Increase Measles Immunization. A Randomized Controlled Trial.
Brief Title: mHealth to Increase Measles Immunization - a Randomized Controlled Trial in Guinea-Bissau
Acronym: mimi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bandim Health Project (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MIMI-01
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Measles
Keywords: mHealth; mobile phones; measles vaccination
MeSH Terms: conditions — Measles

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention)
- Text message (Active Comparator): Subjects in this arm will receive a text message reminder in due time for measles vaccination.
  Interventions: Other: SMS reminder message
- Text message and voice call (Active Comparator): Subjects in this arm will receive a voice call in addition to a text message reminder in due time for measles vaccination.
  Interventions: Other: Voice call + SMS message

INTERVENTIONS:
Other: SMS reminder message
  Arms: Text message
Other: Voice call + SMS message
  Arms: Text message and voice call

SUMMARY:
The question that this project seeks to answer, is whether mobile phones can be used to increase the measles vaccination coverage and timeliness in Guinea-Bissau. The intervention will be evaluated in terms of direct health outcomes and cost/benefit analysis, generating evidence that could help policy makers making informed decisions about implementing mHealth interventions at a national level.

The intervention takes the form of a randomized controlled trial in which text messages (SMS) as well as voice calls are scheduled and delivered to mo thers to remind and encourage them to have their children timely vaccinated against measles. In addition, the messages will include relevant information about opening hours and availability of the measles vaccine at the mothers' local health facilities thus improving coordination. The trial will include three different randomization groups with approx. 350 participants in each group. The first group will receive SMS messages, the second group will receive a voice call in addition to the SMS messages, and the third group is a control group that does not receive any intervention.

Study participants will be enrolled following birth at one of three health centers in different rural regions of Guinea-Bissau. Before the measles vaccine is scheduled to be given, at 9 months of age, mothers will receive the intervention message depending on their assigned randomization group. When the measles vaccine is administered, the child will be registered as having received the measles vaccination.

A follow-up phone interview will be conducted at 12 months of age for all children participating regardless of randomization group and whether or not they received the measles vaccine. All participating children, who at that time still have not received the measles vaccine, will be offered the vaccine at the expense of the project.

ELIGIBILITY:
Inclusion Criteria:

* the mother has access to a cell phone (either her own phone or the phone of a household member)
* the mother lives in the uptake area of the health center.

Exclusion Criteria:

* the mother does not have access to a mobile phone.

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1050 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
MV Coverage at 12 months of age | 12 months of age
  Difference in measles vaccination coverage at 12 months of age between the intervention and the control groups.

SECONDARY OUTCOMES:
Timeliness | At 12 months
  Difference in timeliness of measles vaccines administered, measured as median age of measles vaccinated children.
Average number of visits | At 12 months
  Average number of visits to the health center with the purpose of receiving MV needed before MV is successfully administered.

CONTACTS AND LOCATIONS:
Locations (3):
- Guinea-Bissau (3):
  - Varela Health Center, Varela, Cacheu Region
  - Paunca Health Center, Paunca, Gabú
  - Catio Health Center, Catío, Tombali

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Rossing E, Ravn H, Batista CS, Rodrigues A. MHealth to Improve Measles Immunization in Guinea-Bissau: Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2016 Jul 27;5(3):e158. doi: 10.2196/resprot.5968. PMID 27466046